CLINICAL TRIAL: NCT07378436
Title: A Single-Arm, Single-Center, Open-Label Phase I Clinical Study to Evaluate the Safety, Pharmacokinetics, and Preliminary Efficacy of Autologous Tumor-Reactive T Cells(GK02) Derived From Malignant Ascites Caused by Advanced Solid Tumors
Brief Title: A Clinical Study of GK02 in Malignant Ascites
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing Geekgene Technology Co., LTD (Industry)
Collaborators: Beijing GoBroad Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GK02-GBIIT
Record Dates: First submitted 2026-01-07; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Malignant Ascites Caused by Advanced Solid Tumors
Keywords: Advanced solid tumor; Malignant ascites; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor-reactive T cells-GK02 (Experimental): Treatment with autologous tumor-reactive T cells (GK02) derived from malignant ascites caused by advanced solid tumors.
  Interventions: Drug: GK02

INTERVENTIONS:
Drug: GK02 — Autologous tumor-reactive T cells

SUMMARY:
A single-arm, single-center, open-label clinical study comprising three cohorts, evaluating the safety, preliminary efficacy, and pharmacokinetic/ pharmacodynamic (PK/PD) characteristics of autologous tumor-reactive T cells (GK02) derived from malignant ascites caused by advanced solid tumors.

The trial initially plans to enroll 9 subjects with malignant ascites caused by advanced solid tumors.

DETAILED DESCRIPTION:
To evaluate the safety and preliminary efficacy of an investigational cell therapy, Autologous Tumor-reactive T Cells (GK02) derived from malignant ascites caused by advanced solid tumors.

Following intraperitoneal infusion of GK02, the safety and tolerability of the subjects will be observed, the preliminary effectiveness of the investigational product GK02 in treating malignant ascites will be evaluated, and the pharmacokinetic/pharmacodynamic (PK/PD) characteristics post-administration will be exploratively assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and sign a written informed consent document；
2. At the date of signing ICF, 18 ~75 years old, male or female；
3. Patients with advanced solid tumors confirmed by histology or pathology to have failed at least second-line treatment (treatment failure is defined as progression after treatment or intolerance after treatment), including but not limited to gastric cancer, colorectal cancer, pancreatic cancer, ovarian cancer, etc.；
4. Pathological diagnosis or clinical diagnosis of malignant ascites, and the researcher determines that treatment for malignant ascites is necessary; During screening, the ascites volume was confirmed to be above the medium level by ultrasound (the maximum depth of ascites in the supine position was ≥3.0cm, and the total volume was ≥500ml);
5. ECOG 0-2 points;
6. Adequate organ functions;
7. There are no absolute or relative contraindications for puncture；
8. No peritoneal treatment for malignant ascites has been carried out within 14 days prior to the collection of malignant ascites;
9. Female of childbearing age who have a negative urine pregnancy test during the screening period and agree to take effective contraceptive measures for at least 6 months after perfusion; Male subjects whose partners are fertile must agree to use effective contraceptive methods and avoid sperm donation for at least six months after perfusion.

Exclusion Criteria:

1. Those with a history of severe allergies or allergic reactions to any components of the drugs to be used in this study, including but not limited to NMA-LD drugs, contrast agents and contrast agents used in imaging examinations, excipients such as dimethyl sulfoxide (DMSO) and antibiotics in cell products;
2. Central nervous system (CNS) metastasis is present;
3. Toxicity from previous antitumor therapy did not return to grade 1 or baseline levels (CTCAE version 5.0);
4. Accompanied or prior to interstitial lung disease or interstitial pneumonia;
5. Uncontrolled metabolic disorders, such as those in patients with diabetes (glycated hemoglobin ≥8.5%), or secondary reactions to other non-malignant organ or systemic diseases or cancer, which can lead to higher medical risks and/or uncertainties in survival assessment;
6. An autoimmune disease that is active or has previously suffered from and is likely to recur;
7. Uncontrolled comorbidities include but are not limited to uncontrolled hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg) or any unstable cardiovascular and cerebrovascular diseases that occurred within 6 months prior to treatment enrollment;
8. Ultrasound indicates the separation of peritoneal effusion;
9. Patients with intestinal obstruction;
10. Patients with comorbidities or active autoimmune diseases that require the use of glucocorticoids or other immunosuppressive drugs during the trial period, excluding local transdermal absorption of glucocorticoids (i.e., no more than 5mg/ day of prednisone or equivalent doses of other glucocorticoids);
11. Women who are pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-12-17 (Estimated); Study Completion 2027-12-17 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs | 12 months
  Incidence and severity of AEs, including but not limited to vital signs, physical examination, laboratory tests. All AEs will be classified as Grades 1 through 5 as defined by NCI CTCAE v5.0.
Incidence of DLTs | 28 days
  Number of DLTs (dose limiting toxicities) during the first 28 days after the administrations of GK02 in each cohort.

SECONDARY OUTCOMES:
Changes in the volume of malignant ascites | 12 months
  Change in malignant ascites volume at 28D（day）、2、3、4、5、6、9、12M（month） after GK02 treatment compared to baseline (prior to GK02 infusion).
PuFS | 12 months
  From the first infusion of GK02 to the first paracentesis for ascites drainage or death from any cause.
OS | 12 months
  OS will be assessed from the first GK02 infusion to death from any cause.

OTHER OUTCOMES:
Count of TCR copies | 12 months
  T-cell receptor sequencing (TCR-seq) by obtaining the copy number of the target GK02 T-cell receptors (TCRs) in peripheral blood and malignant ascites： Cmax、Tmax、AUC0-t、AUC0-inf、λz、T1/2.
Concentration of Cytokines | 12 months
  IL-1β、IL-2、IL-4、IL-6、IL-8、IL-10、 IL-12、TGF-b1、IFN-γ and TNF-α
Percentage of Lymphocyte subsets | 12 months
  Total T cells、Th/Ti cells、Ts/Tc cells、NK cells
Proportion of EpCAM + cells | 12 months
  Proportion of EpCAM+ cells among cells

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing GoBroad Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No